CLINICAL TRIAL: NCT05534802
Title: Ulinastatin Improves and Prevents Cardiac Dysfunction Induced by Cardiopulmonary Bypass by Reducing Cardiac Endothelial Permeability
Brief Title: Ulinastatin Improves and Prevents Cardiac Dysfunction Induced by Cardiopulmonary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qin Zhang (Other)
Responsible Party: Sponsor-Investigator, Qin Zhang, phd, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TJ-IRB20220831
Record Dates: First submitted 2022-08-31; First posted 2022-09-10 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Pharmacological Action
Keywords: Cardiac Dysfunction; Cardiac endothelial permeability
MeSH Terms: interventions — urinastatin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: 1. Voluntarily sign the informed consent;
  2. Age ≥18 years old and ≤70 years old;
  3. Patients receiving cardiopulmonary bypass
  4. Patients undergoing heart valve replacement surgery, major vascular surgery, and other cardiac surgery
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment group (Sham Comparator): Cardiac surgery patients undergoing cardiopulmonary bypass are not treated with ulinastatin
  Interventions: Other: saline
- Ulinastatin (Experimental): Cardiac surgery patients undergoing cardiopulmonary bypass are treated with ulinastatin
  Interventions: Drug: Ulinastatin

INTERVENTIONS:
Drug: Ulinastatin — On the basis of conventional treatment, according to the instructions or previous research doses (general anesthesia and tracheal intubation, after cardiopulmonary bypass transfer starts): 10,000 U/kg Ulinastatin (National Medicine Approval No. H19990134, Guangdong Tianpu Biochemical Pharmaceutical Co., Ltd. Co., Ltd., Guangzhou, China) was dissolved in 50 ml of normal saline for 1 hour and pumped through the central vein.
  Arms: Ulinastatin
Other: saline — On the basis of conventional treatment, 50 ml of normal saline for 1 hour and pumped through the central vein.
  Arms: Conventional treatment group

SUMMARY:
This project explores the role and mechanism of ulinastatin in preventing cardiac dysfunction caused by cardiopulmonary bypass by reducing cardiac endothelial permeability through clinical research. Our previous basic research has found that inhibiting the TK/B1R/ARNT/MMP3/iNOS signaling axis in the acute phase of cardiac R/I can reduce the permeability of cardiac endothelial cells, reduce cardiac edema and improve cardiac function (this part has been completed) . This study intends to investigate the effects of ulinastatin on 24-hour cardiac function and prognosis in patients undergoing cardiac surgery undergoing cardiopulmonary bypass (cardiac function, inflammatory indicators, coagulation function, capillary leakage indicators, 28-day survival time, CCU time). At the same time, we observed the dynamic changes of TK/B1R/MMP3 during cardiopulmonary bypass in patients undergoing cardiac surgery and explored its relationship with prognosis, as well as the effect of ulinastatin intervention on TK/B1R/MMP3 before and after cardiopulmonary bypass.

DETAILED DESCRIPTION:
1. Baseline Period Visit 1 (within 24 hours before surgery)

   * Sign informed consent
   * Check inclusion/exclusion criteria
   * Demographic data (sex, age, occupation, etc.)
   * Past medical history (stroke, hypertension, diabetes, dyslipidemia, coronary heart disease, diabetes, etc.) and medication history in the past 3 months
   * Vital signs (temperature, pulse, respiration, blood pressure)
   * Preoperative ECG
   * Preoperative echocardiography
   * Laboratory tests (blood routine, blood glucose, blood lipids, liver and kidney function, myocardial enzymes, blood electrolytes, coagulation function)
   * Concomitant therapy
   * Adverse events
2. Intraoperative cardiopulmonary bypass

   * Record vital signs and various physiological indicators in the operating room.
   * Routinely perform central venous puncture to establish venous access and monitor central venous pressure, and radial artery puncture to monitor invasive arterial pressure.
   * After general anesthesia and endotracheal intubation, routine blood chemistry and arterial blood gas analysis were performed.
   * After collecting the above blood samples for testing, the remaining blood was centrifuged, and the plasma was frozen at -80°C for subsequent testing (levels of CRP, IL-6, IL-10, TNF-α, TK/B1R/MMP3, etc.).
   * Conventional treatment group: On the basis of general anesthesia, the extracorporeal circulation circuit was routinely prefilled. Management of CPB includes blood gas acid-base electrolyte management, anticoagulation management, invasive arterial blood pressure monitoring, MAP in the range of 50-80 mmHg, hematocrit maintained at 20-25%, and non-pulsatile flow rate of 2.0-2.4 L/min/ m2. During cardiopulmonary bypass, the dose of unfractionated heparin for anticoagulation through a central venous catheter is 300-400 U/kg, with additional doses as necessary to achieve and maintain an activated coagulation time (ACT) between 480 and 600 seconds. After isolation from cardiopulmonary bypass, heparin-induced anticoagulation was reversed with protamine. Surgical procedures include coronary artery bypass grafting, heart valve replacement, aortic replacement, etc.
   * Ulinastatin group: On the basis of conventional treatment, administered in accordance with the instructions or previous study doses (general anesthesia with endotracheal intubation, after cardiopulmonary bypass transfer started): 10,000 U/kg Ulinastatin (Guoyao Zhunzi H19990134 , Guangdong Tianpu Biochemical Pharmaceutical Co., Ltd., Guangzhou, China) was dissolved in 50 ml of normal saline for 1 hour through central venous infusion.

   After cardiopulmonary bypass
   * operation time
   * Vital signs (temperature, pulse, respiration, blood pressure)
   * Routine blood chemistry and arterial blood gas analysis
   * Document vasoactive drug use
3. 24 hours, 72 hours, 7 days after surgery

   * Vital signs (temperature, pulse, respiration, blood pressure)
   * Bedside echocardiography
   * Laboratory tests (blood routine, blood sugar, blood lipids, liver and kidney function, myocardial enzymes, coagulation function, etc.)
   * After collecting the above blood samples for testing, the remaining blood is centrifuged, and the plasma is frozen at -80°C for later testing (levels of CRP, IL-6, IL-10, TNF-α, TK/B1R/MMP3, etc.)
   * Capillary leak indicators
   * Document treatment regimen (including vasoactive drug use, etc.)
4. Follow-up period

   * CCU time and total hospital stay
   * 28-day survival status The survival status of the patients was followed up, and the date of death and the cause of death should be recorded in the patients who died.
5. Research Evaluation 1) Main efficacy indicators: cardiac function (echocardiography EF, FS), inflammatory indicators (CRP, IL-6, IL-10, TNF-α), TK/B1R/MMP3 and other levels at 24h, 72h, and 7d after surgery 2) Secondary efficacy indicators: coagulation function, capillary leakage index, 28-day survival rate, CCU time, total hospital stay.
6. Patient Completion/Withdrawal from Study Finish All evaluation data of the patients 28 days after the operation were completely collected and considered as completed cases.

withdraw from the study

Patients will be withdrawn from the study if:

* Patient selection errors
* Intraoperative and postoperative cardiac arrest due to non-CPB causes
* The patient has a drug allergy
* Patient withdraws informed consent
* Any situation in which the investigator believes that the patient should discontinue the study for safety reasons or the patient's interest
* Patient lost to follow-up
* other The date and reason for termination of the study must be recorded on the data collection form. At the time of study termination, patients should be assessed for their final endpoints, in addition to loss to follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent;
2. Age ≥18 years old and ≤70 years old;
3. Patients receiving cardiopulmonary bypass
4. Patients undergoing heart valve replacement surgery, major vascular surgery, and other cardiac surgery

Exclusion Criteria:

1. Severe cardiac insufficiency before surgery (EF<50%, cardiogenic shock);
2. Patients with adverse events during surgery (such as cardiac arrest, etc.);
3. Solid organ or bone marrow transplant recipients;
4. pregnant women;
5. Have a history of allergy to ulinastatin or any of its ingredients;
6. Suffering from autoimmune diseases, tumors, or received high-dose hormones, immunosuppressive drugs, etc. within 2 months;
7. The researcher judges that it is not suitable to participate in this research.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Cardiac function | 24 hours
  Echocardiographic detection
Inflammatory marker | 24 hours
  Detection of CRP
Inflammatory markers | 24 hours
  Detection of IL6
TK/B1R/MMP3 signaling | 24 hours
  Detection levels of tissue kallikrein, B1R and MMP3
POD-postoperative delirium | 7 days
  Assessment Method for the ICU (CAM-ICU

SECONDARY OUTCOMES:
Survival time | 28 days
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liu Y, Wang YL, Zou SH, Sun PF, Zhao Q. Effect of high-dose ulinastatin on the cardiopulmonary bypass-induced inflammatory response in patients undergoing open-heart surgery. Chin Med J (Engl). 2020 Jun 20;133(12):1476-1478. doi: 10.1097/CM9.0000000000000832. No abstract available. PMID 32496303
- [Result] Atal SS, Atal S. Ulinastatin - a newer potential therapeutic option for multiple organ dysfunction syndrome. J Basic Clin Physiol Pharmacol. 2016 Mar;27(2):91-9. doi: 10.1515/jbcpp-2015-0003. PMID 26565549
- [Result] Xu HY, Rong XS, Wang DP, Jiang SY, Zang ZD, Xia W, Zhang F, Yan J. Effect of urinary trypsin inhibitor on inflammatory cytokines and organ function in patients with cardiopulmonary bypass. Eur Rev Med Pharmacol Sci. 2017 May;21(9):2220-2225. PMID 28537661
- Available data/document: Clinical Study Report: 28537661 — https://www.europeanreview.org/article/12702 — Ulinastatin can effectively regulate the inflammatory cytokines and provide protection for organ function during cardiopulmonary bypass surgery, which is conducive to promote the recovery of patients.